CLINICAL TRIAL: NCT03252899
Title: Current Practices of Upper Limb Rehabilitation After Stroke: a Survey Among Stroke Survivors and Therapists
Brief Title: Current Practices of Upper Limb Rehabilitation After Stroke
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/1055
Record Dates: First submitted 2017-07-04; First posted 2017-08-17 (Actual); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Upper Extremity Paresis; Survey
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Therapists: Physiotherapists/occupational therapists experienced in working with stroke patients.
  Interventions: Other: Survey therapists
- Subacute stroke patients: Stroke patients less than 6 months after their stroke suffering from upper limb paresis.
  Interventions: Other: Survey patients
- Chronic stroke patients: Stroke patients more than 6 months after their stroke suffering from upper limb paresis.
  Interventions: Other: Survey patients

INTERVENTIONS:
Other: Survey therapists — A survey was conducted among therapists on upper limb treatment after stroke.
  Groups: Therapists
Other: Survey patients — A survey was conducted among stroke survivors on upper limb treatment after stroke.
  Groups: Chronic stroke patients; Subacute stroke patients

SUMMARY:
A survey was conducted among physiotherapists and occupational therapists working with stroke patients. The survey consisted out of 30 questions enquiring personal information and upper limb specific topics divided in 3 sections: (1) Passive mobilization, (2) Active exercises and (3) Immobilization. The survey took approximately 20 to 30 minutes to complete.

The survey for stroke survivors was divided in seven sections: (1) Personal information (2) Motor recovery of the upper limb and expectations on upper limb recovery; (3) Comfort, pain and quality of life (QoL); (4) Immobilization ; (5) Physiotherapy; (6) Occupational therapy; (7) Nursing (only for patients less than 6 months after stroke). The length to complete the survey was also organized to be achieved in 20 to 30 minutes.

ELIGIBILITY:
Stroke patients

Inclusion Criteria:

* stroke with upper limb paresis

Exclusion Criteria:

* severe language or cognitive problems which make it impossible to complete the survey

Therapists

Inclusion Criteria:

* physiotherapists
* occupational therapists
* experienced in the treatment of stroke patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physiotherapists and occupational therapists Stroke survivors with upper limb impairment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
A questionnaire assessing the current practices of upper limb rehabilitation after stroke | Dec 2016 - March 2017
  To identify the current daily practice in stroke rehabilitation concerning upper limb rehabilitation
A questionnaire assessing the stroke survivors view on upper limb rehabilitation | Dec 2016 - March 2017
  To identify the stroke survivors view on upper limb rehabilitation and understanding the patient needs for that matter.

IPD SHARING:
Plan to Share IPD: No